CLINICAL TRIAL: NCT06052072
Title: Pulmonary Artery DenerVation Clinical Study Using the Gradient Denervation System in Heart Failure Patients With Pulmonary Hypertension Group 2 (PreVail-PH2 Study)
Acronym: PreVail-PH2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gradient Denervation Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-002
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Group 2 Pulmonary Hypertension; Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Prospective, single arm, multi-center, early feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- PADN with Gradient Denervation System (Experimental): Procedure using the Gradient Denervation System to ablate nerves within the pulmonary artery using ultrasonic ablation.
  Interventions: Device: Gradient Denervation System

INTERVENTIONS:
Device: Gradient Denervation System — Pulmonary artery denervation (PADN) procedure using the Gradient Denervation System to ablate nerves within the pulmonary artery using ultrasonic ablation.

SUMMARY:
This early feasibility study is intended to characterize the impact of pulmonary artery denervation on the quality of life in Heart Failure Patients with Group 2 Pulmonary Hypertension

DETAILED DESCRIPTION:
Gradient has developed a novel system for pulmonary artery denervation (PADN) to treat patients with heart failure who also developed pulmonary hypertension (PH). Pulmonary hypertension is frequently associated with left heart failure and is a strong independent predictor of clinical worsening and higher mortality. No therapeutic options are available to treat PH in this selected group of patients with heart failure. The objective is to improve exercise capacity and quality of life by targeting PH in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Heart Failure with EF ≥ 40% (by TTE within last 3 months)
* Mean Pulmonary Artery Pressure (mPAP) >20 mmHg at rest
* Pulmonary Vascular Resistance (PVR) ≥ 3WU at rest
* Pulmonary Capillary Wedge Pressure > 15 mmHg (at rest) or > 18 with passive leg raise
* Cardiac index (CI) ≥ 1.7 L/min/m2
* NYHA Class II or III
* Glomerular Filtration Rate (GFR) ≥ 25 ml/min
* Stable, guideline directed medical treatment, including controlled volume status for a minimum of 3 months prior treatment

Exclusion Criteria:

* Ambulatory with a Life expectancy of < 1 years
* Inability to take dual antiplatelet or anticoagulants, hypersensitivity or allergy to aspirin or clopidogrel
* Unable to tolerate right heart catheterization
* Pulmonary artery aneurysm, moderate or greater PA stenosis or other PA anatomy that would prevent safe or proper use of the study device
* Severe aortic, mitral or pulmonary valve regurgitation
* Tricuspid regurgitation in conjunction with the presence of cirrhosis or congestive hepatopathy
* Clot or Thrombus in any potential target ablation zone (right, left or main pulmonary artery)

Ages: 22 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Device related serious adverse events | Through 30 days post-treatment
  Frequency of SAEs deemed to be related to the investigational device and/or procedure.

SECONDARY OUTCOMES:
Mean change from baseline in Pulmonary Vascular Resistance (woods units) | Measured at 6 months post-treatment
  Calculated mean percent change from baseline

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Northwestern University, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Duke University, Durham, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor College of Medicine, Houston, Texas
  - Houston Methodist, Houston, Texas
  - University of Wisconsin, Madison, Wisconsin
  - Aurora Health, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No